CLINICAL TRIAL: NCT02064400
Title: A Pilot Study of Musculoskeletal Ultrasound Assessment in Patients With Rheumatoid Arthritis
Brief Title: Pilot Study of Ultrasound in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Newcastle University (Other); Wellcome Trust (Other)
Responsible Party: Sponsor
Other Study IDs: NUTH6919
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Ultrasound; Remission; Qualitative
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational study group: Musculoskeletal ultrasound (all patients) and semi-structured patient interview (anticipated maximum 15 patients)
  Interventions: Other: Musculoskeletal Ultrasound; Other: Semi-structured patient interview

INTERVENTIONS:
Other: Musculoskeletal Ultrasound — 7-joint musculoskeletal ultrasound scan
Other: Semi-structured patient interview — Semi-structured patient interview

SUMMARY:
Little is currently known as to the predictive value of ultrasound in guiding the decision to taper drug treatment in patients with stable rheumatoid arthritis, nor the influence that patients' views and opinions regarding their medications may have upon this. In this study, patients with stable rheumatoid arthritis will undergo a simple examination of their joints to look for any swelling or tenderness followed by an ultrasound scan to look for joint inflammation. Half of the patients will also complete an interview to assess their views and opinions of arthritis drug treatment. The study will be completed in a single patient visit - no invasive tests will be performed, and no changes to treatment will be made.

This study is being conducted as part of a Masters degree from Newcastle University. The results of this study will be used to inform the feasibility of inclusion of ultrasound assessment within the design of a future PhD study to investigate potential markers of remission in patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis with symptom onset at least 12 months previously
* Current disease-modifying anti-rheumatic drug (DMARD) therapy or biologic therapy
* Currently stable arthritis defined as no change in DMARD treatment over previous 6 months, and no use of steroids (enteral, parenteral or intra-articular) over previous 6 months

Exclusion Criteria:

* Inability to provide informed consent
* Current or recent (within 4 months) participation within another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary care rheumatology outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Evidence of reliability of intra- and inter-rater ultrasound agreement for power Doppler synovitis score | At recruitment
  Defined as Kappa statistic of at least 0.4.

SECONDARY OUTCOMES:
Qualitative data relating to patients' views and opinions of their arthritis medication | At recruitment
  Based upon data collected by a semi-structured interview approach and analysed using standard qualitative techniques.
Simplified Disease Activity Index (SDAI) | At recruitment
Disease Activity Score in 28 joints (DAS-28) | At recruitment
Disease Activity Score (DAS) | At recruitment

CONTACTS AND LOCATIONS:
Overall Officials: John D Isaacs, PhD, MB BS, Principal Investigator — Newcastle University
Locations (1):
- Musculoskeletal Outpatient Department, Freeman Hospital, Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] Baker KF, Isaacs JD, Thompson B. "Living a normal life": a qualitative study of patients' views of medication withdrawal in rheumatoid arthritis. BMC Rheumatol. 2019 Jun 13;3:2. doi: 10.1186/s41927-019-0070-y. eCollection 2019. PMID 31225429